CLINICAL TRIAL: NCT02341482
Title: A Phase 1, Open-label, Fixed-sequence Study To Estimate The Effects Of Multiple-dose Administration Of Itraconazole On The Pharmacokinetics Of Pf 04958242 In Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of PF-04958242 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1701021; DDI (Other: Alias Study Number)
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Results first posted 2016-06-30 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Healthy
Keywords: Itraconazole; Healthy Volunteers; Drug-drug interaction; PF-04958242
MeSH Terms: interventions — PF-04958242; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-04958242 and itraconazole (Experimental): PF-04958242 will be provided in a capsule. Participants will receive a 0.10 mg loading dose of PF-04958242 twice daily (BID) on Day 1 then 0.025 mg BID on Day 2-Day 16, with the last dose occurring in the morning on Day 17.
  Itraconazole will be provided as a solution starting on Day 4. On Day 4, a 200 mg dose of itraconazole will be administered approximately 1 hour before PF-04958242 morning administration and for 13 additional days (Day 4-Day 17).
  Interventions: Drug: PF-04958242; Drug: Itraconazole

INTERVENTIONS:
Drug: PF-04958242 — Administered as specified in the treatment arm
Drug: Itraconazole — Administered as specified in the treatment arm

SUMMARY:
The purpose of the current study is to characterize the pharmacokinetic (PK) profile of PF 04958242 when co administered with a strong cytochrome P450 3A4 (CYP3A4) inhibitor.

DETAILED DESCRIPTION:
This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

-Healthy male subjects and female subjects of non childbearing with a Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >55 kg (121 lbs).

Key Exclusion Criteria:

* Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat, if deemed necessary:

  * Aspartate transaminase (AST)/serum glutamic oxaloacetic transminase (SGOT) or alanine transaminase (ALT)/serum glutamic pyruvic transminase (SGPT) >=1 x upper limit of normal (ULN);
  * Total bilirubin >=1.5 x ULN; subjects with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is <= ULN.
* Subjects with epilepsy, or history of epilepsy, or conditions that lower seizure threshold, seizures of any etiology (including substance or drug withdrawal), or who have increased risk of seizures as evidenced by self reported history of electroencephalogram (EEG) with epileptiform activity. Subjects with a history of childhood seizures and history of head trauma with loss of consciousness requiring hospitalization overnight will be excluded as well.
* Subjects who had a history of allergy or intolerance to azole antifungal drugs.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: PF-04958242 0.10 milligram (mg) loading dose was administered orally twice daily (BID) on Day 1. Each participant was given 2 daily doses of PF-04958242 (0.025 mg) orally for 16 subsequent days (Day 2 to Day 17), with the last dose occurring in the morning of Day 17. On Day 4, a 200 mg dose of itraconazole was administered orally approximately 1 hour before PF-04958242 morning administration and for 13 additional days (Day 4 to Day 17), once daily (QD).
Period: Overall Study
Arm/Group | All Subjects
Started | 13
Completed | 12
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: PF-04958242 0.10 mg loading dose was administered orally BID on Day 1. Each participant was given 2 daily doses of PF-04958242 (0.025 mg) orally for 16 subsequent days (Day 2 to Day 17), with the last dose occurring in the morning of Day 17. On Day 4, a 200 mg dose of itraconazole was administered orally approximately 1 hour before PF-04958242 morning administration and for 13 additional days (Day 4 to Day 17), QD.
Arm/Group | All Subjects
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Profile From Time 0 to Time Tau, the Dosing Interval, Where Tau = 12 Hours (AUCtau) of PF-04958242
Description: AUCtau = area under the concentration-time profile from time 0 to time tau, the dosing interval, where tau = 12 hours. Collected at Day 3 for PF-04958242 0.025 mg Arm and Day 17 for PF-04958242 0.025 mg + itraconazole 200 mg Arm.
Time Frame: Day 1 (0,1.5,12,13.5 hours post-dose), Day 2 (0,1.5,12,13.5 hours post-dose), Day 3 (0,0.5,1,1.5,2,3,4,6,8,12 hours post-dose), Day 4, Day 7, Day 10, Day 13, Day 16, Day 17 (0,0.5,1,1.5,2,3,4,5,6,8,12 hours post-dose) Day 18, Day 19, Day 20, Day 21
Population: The PK analysis population included all participants enrolled and treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hours per milliliter pg*h/mL
Groups:
- PF-04958242 0.025 mg: All participants who received PF-04958242 0.025 mg BID orally.
- PF-04958242 0.025 mg + Itraconazole 200 mg: All participants who received PF-04958242 0.025 mg BID combined with Itraconazole 200 mg QD orally.
Arm/Group | PF-04958242 0.025 mg | PF-04958242 0.025 mg + Itraconazole 200 mg
Number analyzed (Participants) | 13 | 12
picogram*hours per milliliter pg*h/mL | 4242 (30) | 4073 (25)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04958242
Description: Collected at Day 3 for PF-04958242 0.025 mg Arm and Day 17 for PF-04958242 0.025 mg + itraconazole 200 mg Arm.
Time Frame: as for outcome 1
Population: All enrolled participants treated who received at least 1 dose of PF-04958242 and had at least 1 measureable concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PF-04958242 0.025 mg | PF-04958242 0.025 mg + Itraconazole 200 mg
Number analyzed (Participants) | 13 | 12
pg/mL | 553.4 (27) | 541.6 (20)

3. Secondary Outcome: Time for Cmax (Tmax) of PF-04958242
Description: Collected at Day 3 for PF-04958242 0.025 mg Arm and Day 17 for PF-04958242 0.025 mg + itraconazole 200 mg Arm.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04958242 0.025 mg | PF-04958242 0.025 mg + Itraconazole 200 mg
Number analyzed (Participants) | 13 | 12
hours | 1.50 [1.00 to 1.52] | 1.50 [1.00 to 2.00]

4. Secondary Outcome: Lowest Concentration Observed During the Dosing Interval (Cmin) of PF-04958242
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PF-04958242 0.025 mg | PF-04958242 0.025 mg + Itraconazole 200 mg
Number analyzed (Participants) | 13 | 12
pg/mL | 256.5 (35) | 238.2 (30)

5. Secondary Outcome: Predose Concentration (Ctrough) of PF-04958242
Time Frame: 0 hour at Day 1, Day 2, Day 3, Day 4, Day 7, Day 10, Day 13, Day 16, and Day 17 (pre-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PF-04958242 0.025 mg | PF-04958242 0.025 mg + Itraconazole 200 mg
Number analyzed (Participants) | 13 | 12
pg/mL | 289.3 (37) | 255.0 (29)

6. Secondary Outcome: Apparent Oral Clearance (CL/F) of PF-04958242
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Collected at Day 3 for PF-04958242 0.025 mg Arm and Day 17 for PF-04958242 0.025 mg + itraconazole 200 mg Arm.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per minute (mL/min)
Arm/Group | PF-04958242 0.025 mg | PF-04958242 0.025 mg + Itraconazole 200 mg
Number analyzed (Participants) | 13 | 12
milliliters per minute (mL/min) | 98.25 (30) | 102.3 (25)

7. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Measurements
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, mean corpuscular volume [MCV], mean corpuscular hemoglobin [MCH], mean corpuscular hemoglobin concentration [MCHC], platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen [BUN], creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, alkaline phosphatase, uric acid, albumin, and total protein; urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin and microscopy [if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase]); others (follicle stimulating hormone [FSH], urine cotinine, and urine drug screening).
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 13
participants | 1

8. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Criteria of Potential Clinical Concern
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: supine/sitting pulse rate more than (<)40 or less than (>)120 beats per minute (bpm); systolic blood pressure (SBP) more than or equal to (>=)30 millimeters of mercury (mm Hg) change from baseline in same posture or SBP <90 mm Hg, diastolic blood pressure (DBP) >=20 mm Hg change from baseline in same posture or DBP <50 mm Hg. IFB = increase from baseline; DFB = decrease from baseline.
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 13
participants
  Supine SBP <90 mmHg | 0
  Supine DBP <50 mmHg | 0
  Supine Pulse Rate <40 BPM | 0
  Supine Pulse Rate >120 BPM | 0
  Supine SBP >=30 mmHg IFB | 2
  Supine DBP >=20 mmHg IFB | 1
  Supine SBP >=30 mmHg DFB | 0
  Supine DBP >=20 mmHg DFB | 0

9. Secondary Outcome: Number of Participants With Electrocardiogram Data Meeting Criteria of Potential Clinical Concern
Description: Electrocardiogram (ECG) parameters included time from ECG Q wave to the end of the T wave corresponding to electrical systole (QT) interval, beginning of the P wave until the beginning of the QRS complex (PR) interval, time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS) interval, QT interval corrected for heart rate (QTc) interval, and corrected QT interval using Fridericia's formula (QTcF). Criteria for ECG changes meeting potential clinical concern included: PR interval >=300 milliseconds (msec) or >=25% increase when baseline is >200 msec and >=50% increase when baseline is less than or equal to (=<)200 msec; QRS interval >=140 msec or >=50% increase from baseline; and QTcF >=450 to <480, 480 to <500 and >=500 msec or >=30 to 60 msec increase and also >=60 msec increase. The number of participants with potentially clinically significant ECG findings at any visit were reported.
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 13
participants | 0

10. Secondary Outcome: Number of Participants With Significant Change in Neurological Examination From Previous Examination
Description: The extended neurological examination, performed by a board certified neurologist, included observations for cerebellar (intention) tremor and for non-cerebellar tremors (eg, resting or positional), finger, nose, heel, shin, Romberg, tandem walking, positional and gaze evoked nystagmus, reflexes, muscle strength, cranial nerves, sensory function of upper and lower extremities. The brief neurological examination included an assessment of motor and sensory function, cranial nerves, reflexes, non-cerebellar tremor (eg, resting or positional) and cerebellar function. The assessment of cerebellar function were complemented by the Scale for Assessment and Rating of Ataxia (SARA).
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 13
participants | 0

11. Secondary Outcome: Number of Participants With Significant Change in Physical Examination From Previous Examination
Description: A full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The brief physical examination focused on general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms.
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 13
participants | 0

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to 28 days after last study drug administration
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Groups:
- PF-04958242 0.1 mg: All participants who received PF-04958242 0.1 mg BID orally.
Arm/Group | PF-04958242 0.025 mg | PF-04958242 0.025 mg + Itraconazole 200 mg | PF-04958242 0.1 mg
Number analyzed (Participants) | 13 | 13 | 13
participants
  AEs | 2 | 7 | 1
  SAEs | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Positive Response to Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment [C-CASA]) is an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced the following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3)("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7)("Yes" on "Has participant engaged in non-suicidal self-injurious behavior").
Time Frame: Baseline up to Day 21
Population: The safety analysis population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 13
participants | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug.
Groups:
- PF-04958242 0.025 mg Combined With Itraconazole 200 mg: All participants who received PF-04958242 0.025 mg combined with itraconazole 200 mg orally.
Arm/Group | PF-04958242 0.1 mg | PF-04958242 0.025 mg | PF-04958242 0.025 mg Combined With Itraconazole 200 mg
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 2/13 | 7/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04958242 0.1 mg (N=13) | PF-04958242 0.025 mg (N=13) | PF-04958242 0.025 mg Combined With Itraconazole 200 mg (N=13)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Drug intolerance (General disorders) | 0 | 0 | 1
Fat tissue increased (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 2
Penile swelling (Reproductive system and breast disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No